CLINICAL TRIAL: NCT03677726
Title: Improving Sleep Continuity Through Mindfulness Training for Better Cognitive Ageing.
Acronym: MIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017/2830
Record Dates: First submitted 2018-08-13; First posted 2018-09-19 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Sleep Initiation and Maintenance Disorders; Cognitive Aging
Keywords: Insomnia; Cognitive aging; Mindfulness
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either a Mindfulness-based Therapy for Insomnia (MBTI) or a Sleep Hygiene Education Program (SHEP). The intervention is for 8 weeks. Measures will be administered prior to and on completion of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Therapy for Insomnia (Experimental): The mindfulness-based intervention consists of eight 2-hour sessions covering various mindfulness techniques (e.g. mindfulness of breath, body and movement, senses and informal practice, and empathy and compassion) that pertain to people with sleep problems and insomnia. Participants will be provided handouts for the information covered during these talks and discussions.
  Interventions: Behavioral: Mindfulness Based Therapy for Insomnia
- Sleep Hygiene Education Exercise Program (Active Comparator): The Sleep Hygiene Education and Exercise Program has known relationships with good sleep quality. It will comprise of eight weekly 2-hour sessions. Each session will introduce a concept related to sleep and sleep hygiene. The facilitator will provide the theory and rationale behind the concept, and encourage participants to share and discuss their experiences related to the concept. The session will end with the participants evaluating how to implement the specific concept in their daily lives, and its potential implications for their sleep. Participants will be provided with a manual that outlines the concept and how they intend to apply it to their daily lives.
  Interventions: Other: Sleep Hygiene Education Exercise Program

INTERVENTIONS:
Behavioral: Mindfulness Based Therapy for Insomnia — The mindfulness-based intervention consists of eight 2-hour sessions covering various mindfulness techniques (e.g. mindfulness of breath, body and movement, senses and informal practice, and empathy and compassion) that pertain to people with sleep problems and insomnia. Participants will be provided handouts for the information covered during these talks and discussions.
  Other Names: MBTI
  Arms: Mindfulness Based Therapy for Insomnia
Other: Sleep Hygiene Education Exercise Program — The Sleep Hygiene Education and Exercise Program has known relationships with good sleep quality. It will comprise 8 weekly 2-hour sessions. Each session will introduce a concept related to sleep and sleep hygiene. The facilitator will provide the theory and rationale behind the concept, and encourage participants to share and discuss their experiences related to the concept. The session will end with the participants evaluating how to implement the specific concept in their daily lives, and its potential implications for their sleep. Participants will be provided with a manual that outlines the concept and how they intend to apply it to their daily lives.
  Other Names: SHEEP
  Arms: Sleep Hygiene Education Exercise Program

SUMMARY:
Poor sleep quality is a known risk factor for cognitive decline in the elderly. Hearteningly, sleep is also a prime target for behavioral modification. In this study, the investigators propose to test mindfulness-based training (MBT) as an intervention to improve sleep quality by reducing sleep fragmentation, and hypothesize that these improvements will mediate the beneficial effects of MBT on sustained and executive attention. MBT consists of a suite of techniques aimed at enhancing awareness and acceptance of one's internal (e.g., thoughts and feelings) and external experiences in the present moment. Learning these techniques has been shown to improve sleep quality in patients with primary insomnia, and in other conditions associated with sleep disturbance. There is also increasing evidence that mindfulness training enhances multiple facets of cognition, including components of attention. In this study, the investigators will recruit 120 participants in a randomized controlled design, with 60 participants receiving MBT, and 60 receiving a sleep hygiene education and exercise program (SHEEP). Each intervention will last 8 weeks. Before and after the intervention, the investigators will collect objective and subjective measures of sleep quality, resting-state and task-related functional magnetic resonance imaging scans, and performance on standard laboratory tests of attention. The investigators hypothesize that, relative to SHE, MBT will result in significantly greater improvements in sleep quality and attentional metrics. They also predict that the cognitive changes will be mediated by the changes in sleep quality. If a positive result is found, this would indicate the use of MBT as a cost-effective behavioral intervention to stabilize or even improve cognition in the elderly, thus reducing the risk of dementia in this vulnerable population.

DETAILED DESCRIPTION:
Cognitive decline in the elderly is a rapidly growing concern in Singapore and other developed Asian nations. Among the major but understudied factors that may exacerbate this decline is poor sleep quality. Targeting sleep to decelerate or even reverse age-related cognitive decline may represent a low-cost, high-return solution to a widespread societal problem.

To accomplish this goal, the investigators propose to test mindfulness-based training (MBT) as an intervention to improve sleep quality and cognition.

In this pilot grant, the investigators will study a group of participants (N = 120) in a randomized controlled design pitting MBT (N =60) against sleep hygiene education (SHEEP, N = 60).

Hypothesis 1: MBT will lead to significantly greater improvements in sustained and executive attention relative to SHEEP (measured both behaviorally and using functional magnetic resonance imaging).

Hypothesis 2: Cognitive outcomes will be mediated by improvements in subjective and objective sleep quality.

Good sleep is critical for cognition at all ages, and especially in the elderly

Adequate sleep is important for optimal cognitive function across the lifespan. Although the association between sleep and cognitive function is bi-directional, alterations in sleep frequently occur prior to the appearance of cognitive symptoms in Alzheimer's Disease (AD). Almost 50% of older adults report at least one sleep problem, and there is growing evidence that sleep complaints and disturbances might have negative effects on cognition.

Retired older adults have the freedom to sleep ad libitum but this benefit is offset by age-associated changes in sleep such as poorer subjective quality, increased fragmentation and/or altered macrostructure. Although sleep duration is the measure that has received the most attention, there is accumulating evidence that sleep quality (Blackwell et al., 2014) and sleep fragmentation in particular, can have deleterious effects on brain structure and cognition. A change in sleep pattern in late adulthood can foreshadow cognitive decline, perhaps as a result of accumulation of neurotoxic substances that are normally cleared during sleep.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 50 to 80
2. English-speaking
3. Mini-Mental State Examination Score ≥ 26
4. Montreal Cognitive Assessment Score ≥ 23

At least one of the following sleep difficulties are expressed:

(i) average reported sleep latency of more than 30 minutes

(ii) average wakefulness after sleep onset of more than 30 minutes

(iii) sleep efficiency or total sleep time of less than 6.5 hours

and/or

(iv) also a cut off in the PSQI>/=5

Exclusion Criteria:

1. Presence of major neurological conditions such as epilepsy, stroke, Parkinson's Disease and/or brain injury
2. Presence of major psychiatric conditions such as major depression or schizophrenia
3. Unsuitability for fMRI scanning (e.g. pacemakers, metallic implants, claustrophobia)
4. Unable to give independent consent or no consent available

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Change in Subjective measures of Sleep quality: Pittsburgh Sleep Quality Index Score | Up to one month
  Pittsburgh Sleep Quality Index Score (PSQI) is a 19-item self-rated questionnaire for evaluating subjective sleep quality over the previous month. The PSQI has a sensitivity of 89.6% and specificity of 86.5% for identifying cases with sleep disorder, using a cut-off score of 5.
  The first 4 items are open questions, whereas items 5 to 19 are rated on a 4-point Likert scale. Individual items scores yield 7 components. A total score, ranging from 0 to 21, is obtained by adding the 7 component scores. A score of 5 and above suggests poor sleep quality. A decrease in PSQI score following intervention would reflect and improvement of sleep quality.
Polysomnography: objective changes in sleep onset latency (SOL) | One night
  Polysomnography is a multi-parametric test used in the study of sleep and as a diagnostic tool in sleep medicine. PSG is a comprehensive recording of bio-physiological changes that occur during sleep. It will be performed at night, at the convenience of the participants' home. PSG monitors many body functions including brain, eye movements, muscle activity or skeletal muscle activation and heart rhythm during sleep. The investigators will use a Somnimedics PSG kit. Sleep onset latency reflects the amount of time it takes to participants to fall asleep from the moment they go to bed in the evening, so higher SOL are indicative of poor sleep quality.
  This objective measure of participants sleep onset latency will judge sleep quality against the subjective measures obtained through the sleep questionnaires.
Actiwatch: objective changes in sleep onset latency (SOL) | One week
  Wrist-worn actigraphy is a convenient and reliable way to monitor sleep. It will be performed using research-grade, wrist-worn accelerometers that are calibrated to detect sleep by inferring from movement patterns. The systems used in this proposal (Philips Respironics AW-2 or Spectrum) has been calibrated against PSG. Sleep onset latency reflects the amount of time it takes to participants to fall asleep from the moment they go to bed in the evening, on average over seven nights of recording.
  This objective measure of participants sleep onset latency will judge sleep quality against the subjective measures obtained through the sleep questionnaires.
Polysomnography: objective changes in wake after sleep onset (WASO) | One night
  In addition to Sleep Onset Latency (Primary outcome 2), a second objective measure of sleep quality is extracted from the polysomnography recording: periods of wakefulness occurring after defined sleep onset. WASO is calculated by taking into account the total time spent in bed, minus sleep latency and minus total sleep time. High WASO scores reflect low sleep continuity and poor sleep quality.
  This second measure of participants sleep will judge sleep quality against the subjective measures obtained through the sleep questionnaires.
Actiwatch: objective changes in wake after sleep onset (WASO) | One week
  As with measures from PSG, in addition to Sleep Onset Latency (Primary outcome 3), a second objective measure of sleep quality is extracted from the Actiwatch recording: periods of wakefulness occurring after defined sleep onset. WASO is calculated by taking into account the total time spent in bed, minus sleep latency and minus total sleep time, averaged over seven consecutive nights.
  This second measure of participants sleep will judge sleep quality against the subjective measures obtained through the sleep questionnaires.
Change in Subjective measures of Sleep quality: Insomnia Severity Index | Past two weeks
  Insomnia Severity Index (ISI) evaluates an individual's level of tendency for insomnia on a 7-item questionnaire, scoring in total from 0 to 28. Scores above 15 indicates moderate severity of clinical insomnia while scores above 22 are indicative of severe clinical insomnia. ISI internal consistency was excellent for population samples both in the community and clinical samples as well, (Cronbach α of 0.90 and 0.91 respectively).
Change in Cognitive and Attention tasks performance (CANTAB: Reaction time task) | Up to 10 minutes
  Reaction time task (RTI) provides assays of motor and mental response speeds, as well as measures of movement time, reaction time and response accuracy. Primary outcome: reaction times. Lower reaction times are indicative of better performance.
Change in Cognitive and Attention tasks performance (CANTAB: Rapid Visual Information Processing primary outcome) | Up to 10 minutes
  Rapid Visual Information Processing (RVP) is a sensitive tool for assessment of sustained attention. Primary outcomes: median response latency. Lower scores in this measure reflect better sustained attention.
Change in Cognitive and Attention tasks performance (CANTAB: Paired Associate Learning) | Up to 10 minutes
  Paired Associate Learning (PAL) assesses visual memory and new learning, and is a sensitive tool for accurate assessment of episodic memory. Primary outcome: accuracy on first trials memory score
Change in Cognitive and Attention tasks performance (CANTAB: Spatial Working Memory) | Up to 10 minutes
  Spatial Working Memory (SWM) requires retention and manipulation of visuospatial information. This test has notable executive function demands, and measures strategy use as well as errors. Primary outcome: number of errors.
Change in Cognitive and Attention tasks performance (CANTAB: Stocking of Cambridge) | Up to 10 minutes
  Stocking of Cambridge (SOC) assesses spatial planning and requires individuals to use problem-solving strategies to match two sets of stimuli. Primary outcome: number of problems solved on first choice.

SECONDARY OUTCOMES:
Imaging measures (structural): change in orbitofrontal cortex volume | 6 minutes
  Structural and MRI brain scans will be used to assess the change in the volume of orbitofrontal cortex (OFC) - the key region that is both consistently altered by mindfulness meditation, leading to an increase in volume, and implicated in sleep pathology. Participants will have their baseline fMRI scan at least 1-week before the start of their participation in the intervention and after the end of the intervention.
Change in functional imaging measures: Resting state and Inscape | 10 minutes
  During two rsfMRI scans, subjects are imaged over several minutes while their eyes are open, but without performing any explicit task. It has been recognized that a person's brain activity at rest contains a rich source of information about their brain function. One of the resting state scan will show only a fixation cross on the screen (resting state), and the second one (Inscape) will show a short video developed in order to minimize the cognitive processing involved while decreasing head movement and sleepiness in the scanner.
  These data are typically extracted by decomposing the time-varying signal during resting periods into independent, intrinsically connected networks. The investigators propose to use traditional connectivity analysis as well as a newer method: graph theory analysis Measure will be increase of task ready state in Dynamic Functional Connectivity, as previous literature suggested that this is positively linked with mindfulness predisposition.
Change in functional imaging measures: Breath counting task | 10 minutes
  Main measure is change in cortical activity during sustained attention task, before and after intervention.
  Similar analysis to the resting-state fMRI scans will be conducted to determine the change in Default Mode Network (DMN) and Executive Control Network (ECN) connectivity and anti-correlation between DMN and task-positive networks.
Change in functional imaging measures: Letting go practice | 10 minutes
  Change in cortical connectivity while performing a Letting go practice in the scanner. Analysis are similar to the resting state and breath counting task (outcomes 13 and 14).
Change in Cognitive and Attention tasks performance (CANTAB: Emotion Recognition Task) | Up to 10 minutes
  Emotion Recognition Task: ERT assesses social cognition and measures the ability of the subject to identify emotions in facial expressions. Secondary outcomes: Accuracy and Reaction times.
Change in Cognitive and Attention tasks performance (CANTAB: Verbal Recognition Memory) | Up to 10 minutes
  Verbal Recognition Memory: RM measures the ability to encode and subsequently retrieve verbal information. Secondary outcomes: number of correct-incorrect responses. Higher scores are indicative of better verbal recognition memory.
Change in Cognitive and Attention tasks performance (CANTAB: Rapid Visual Information Processing) | Up to 10 minutes
  Rapid Visual Information Processing: RVP is a sensitive tool for assessment of sustained attention. Secondary outcomes: A prime. Higher scores in this measure reflects better performance.
Behavioral Breath counting task: Errors | 20 minutes
  BCT is a behavioural measure of trait mindfulness found to be reliable and correlated with self-report mindfulness. Outcome measure: number of errors.
Behavioral Breath counting task: Accuracy | 20 minutes
  BCT is a behavioural measure of trait mindfulness found to be reliable and correlated with self-report mindfulness. Outcome measure: accuracy and number of miscounts and resets.
Pen and Pencil cognitive test: Colour Trails A and B | Up to 30 minutes
  Widely used instrument in neuropsychological assessment to measure for speed of cognitive processing and executive functioning. The direct score of both parts A and B are represented by the time taken to complete each task.
Pen and Pencil cognitive test: IQ Advances Progressive Matrices I and II | Up to 30 minutes
  This test is a nonverbal group test typically used in educational settings. It is a 60-item test used in measuring abstract reasoning and regarded as a non-verbal estimate of fluid intelligence.
Five Facet Mindfulness Questionnaire (FFMQ) | Past one month
  This 39-item instrument is based on a factor analytic study of five independently developed mindfulness questionnaires. The analysis yielded five factors that appear to represent elements of mindfulness as it is currently conceptualized. The five facets are observing (8 items), describing (8 items), acting with awareness (8 items), non-judging of inner experience (8 items), and non-reactivity to inner experience (7 items). Scores for each subscales are calculated as the mean of the items, ranging from 1 to 5. Total FFMQ score is the mean of all the subscales, ranging 1-5.
Change in Subjective measures of Sleep quality: Dysfunctional Beliefs and Attitudes about Sleep | Past one month
  Dysfunctional Beliefs and Attitudes about Sleep (DBAS) is a 30-item self reported questionnaire to measure people's beliefs and attitudes about their personal sleep situations. Items are ranked from 0, strongly disagree, to 10, strongly agree. Total score is mean of all questions, with a higher score representing more dysfunctional beliefs and attitude about sleep.
Change in Subjective measures of Sleep quality: Pre-Sleep Arousal, | Past one month
  Pre-Sleep Arousal, PSA is a 16-item self report questionnaire having both cognitive and somatic dimensions of arousal. Scores on each subscale range from 8-40 (sum of individual answers); high scores on both subscale indicate more arousal. The Cronbach alpha of this scale was .88 and test-retest reliability is .72.
Change in Subjective measures about mood, anxiety and quality of life: State Trait Anxiety Inventory | Past year
  State Trait Anxiety Inventory (STAI) has 40 items, 20 items allocated to each of the State-Anxiety (questions 1-8) and Trait-Anxiety (questions 9-16) subscales, each ranging from 20 to 80. It is a self-report questionnaires to indicate the presence and severity of current symptoms of anxiety and a generalized propensity to be anxious. Higher scores are positively correlated with higher levels of anxiety.
Change in Subjective measures about mood, anxiety and quality of life: Beck's Depression Inventory, | Up to last year
  Beck's Depression Inventory (BDI-II) is a 21- item questionnaire that evaluates the severity of depressive mood states. Each item is rated between 0 (no symptom impact) and 3 (maximum symptom impact) with a maximum score of 63. Two domains are evaluated: the cognitive-affective (questions 1-13, ranging from 0 to 39) and somatic domains (questions 14-21, ranging from 0 to 24). Higher scores in both subscales represent lower mood and more depressive symptoms.
Change in Subjective measures about mood, anxiety and quality of life: Short-Form 36 | Up to last year
  Short-Form 36 (SF-36) is a 36-item self-report survey of health, including physical and mental health, with 8 scaled scores, each ranging from a minimum of 0 to max 100. Total score is the mean of all the subscales.
  Physical functioning : 10 items; Role functioning/physical : 4 items; Role emotional: 3 items; Energy/fatigue: 4 items; Mental Health: 5 items; Social functioning: 2 items; Body pain: 2 items; General health : 5 items; Reported health transition: 1 item.
Polysomnography: objective changes in total sleep time (TST) | One night
  Polysomnography is a multi-parametric test used in the study of sleep and as a diagnostic tool in sleep medicine. It will be performed at night, at the convenience of the participants' home. Total sleep time reflects the amount of time participants were effectively sleeping while in bed, without periods of wakefulness.
  This objective measure of participants total sleep time will judge sleep quality against the subjective measures obtained through the sleep questionnaires.
Actiwatch: objective changes in total sleep time (TST) | One week
  Wrist-worn actigraphy is a convenient and reliable way to monitor sleep. Total sleep time reflects the amount of time participants were effectively sleeping while in bed, without periods of wakefulness, on average over seven nights of recording.
  This objective measure of participants total sleep time will judge sleep quality against the subjective measures obtained through the sleep questionnaires.
Change in oxygen levels during sleep | One night
  A Pulse Oximetry (SPO device from Somnotouch RESP, SomnoMedics) will be clipped at the end of participants' finger overnight together with the PSG recording, pre and post intervention, to measure peripheral capillary oxygen saturation changes.
  When compared with PSG and Actiwatch measures, oxygen levels can provide additional information about sleep quality. A decrease in oxygen level is often linked to sleep disorders like obstructive sleep apnea.
Heart rate during sleep | One night
  The Pulse Oximetry used for measuring oxygen levels for outcome 31 can also provide information about heart rate during sleep. Heart rate will be recorded for a full night before and after the intervention, together with PSG. Heart rate for adults during sleep varies widely across individuals, usually between 40-100 beats per minute.

CONTACTS AND LOCATIONS:
Overall Officials: Kinjal Doshi, Principal Investigator — Singapore General Hospital; Julian Lim, Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided
Preliminary data to inform design of future studies.

REFERENCES:
- [Background] Lim J, Teng J, Patanaik A, Tandi J, Massar SAA. Dynamic functional connectivity markers of objective trait mindfulness. Neuroimage. 2018 Aug 1;176:193-202. doi: 10.1016/j.neuroimage.2018.04.056. Epub 2018 Apr 27. PMID 29709625
- [Background] F Wong K, A A Massar S, Chee MWL, Lim J. Towards an Objective Measure of Mindfulness: Replicating and Extending the Features of the Breath-Counting Task. Mindfulness (N Y). 2018;9(5):1402-1410. doi: 10.1007/s12671-017-0880-1. Epub 2018 Jan 22. PMID 30294387
- [Background] Blackwell T, Yaffe K, Laffan A, Ancoli-Israel S, Redline S, Ensrud KE, Song Y, Stone KL; Osteoporotic Fractures in Men (MrOS) Study Group. Associations of objectively and subjectively measured sleep quality with subsequent cognitive decline in older community-dwelling men: the MrOS sleep study. Sleep. 2014 Apr 1;37(4):655-63. doi: 10.5665/sleep.3562. PMID 24899757
- [Background] Lim J, Dinges DF. A meta-analysis of the impact of short-term sleep deprivation on cognitive variables. Psychol Bull. 2010 May;136(3):375-89. doi: 10.1037/a0018883. PMID 20438143
- [Background] Ju YE, Lucey BP, Holtzman DM. Sleep and Alzheimer disease pathology--a bidirectional relationship. Nat Rev Neurol. 2014 Feb;10(2):115-9. doi: 10.1038/nrneurol.2013.269. Epub 2013 Dec 24. PMID 24366271
- [Background] Lim AS, Kowgier M, Yu L, Buchman AS, Bennett DA. Sleep Fragmentation and the Risk of Incident Alzheimer's Disease and Cognitive Decline in Older Persons. Sleep. 2013 Jul 1;36(7):1027-1032. doi: 10.5665/sleep.2802. PMID 23814339
- [Derived] Shaif NAS, Doshi K, Lim J. Effects of mindfulness-based therapy for insomnia and a sleep hygiene/exercise programme on subjective-objective sleep discrepancy in older adults with sleep disturbances: Exploratory secondary analysis of a randomised clinical trial. J Sleep Res. 2022 Dec;31(6):e13700. doi: 10.1111/jsr.13700. Epub 2022 Jul 27. PMID 35896519
- [Derived] Perini F, Wong KF, Lin J, Hassirim Z, Ong JL, Lo J, Ong JC, Doshi K, Lim J. Mindfulness-based therapy for insomnia for older adults with sleep difficulties: a randomized clinical trial. Psychol Med. 2023 Feb;53(3):1038-1048. doi: 10.1017/S0033291721002476. Epub 2021 Jul 1. PMID 34193328